CLINICAL TRIAL: NCT02664805
Title: A Phase 2a, Proof of Concept Trial, Testing Twice Daily Applications of LEO 124249 Ointment in the Treatment of Chronic Hand Eczema
Brief Title: Proof of Concept, Twice Daily Applications of LEO 124249 Ointment in the Treatment of Chronic Hand Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0133-1180; 2015-002079-11 (EudraCT Number)
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2018-03

CONDITIONS: Hand Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 124249 ointment (Active Comparator): Twice daily cutaneous application for 8 weeks
  Interventions: Drug: LEO 124249 ointment
- LEO 124249 ointment vehicle (Placebo Comparator): Twice daily cutaneous application for 8 weeks
  Interventions: Drug: LEO 124249 ointment vehicle

INTERVENTIONS:
Drug: LEO 124249 ointment — Ointment
  Arms: LEO 124249 ointment
Drug: LEO 124249 ointment vehicle — Ointment vehicle
  Arms: LEO 124249 ointment vehicle

SUMMARY:
To compare the efficacy of twice daily applications of LEO 124249 ointment with LEO 124249 ointment vehicle for up to 8 weeks in the treatment of subjects with chronic hand eczema.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic hand eczema with or without atopic etiology/background with a history of not adequately controlled disease activity with cutaneously applied steroid
* Physician's Global Assessment of disease severity graded as at least mild at Visit 1
* In overall good health including well controlled diseases

Exclusion Criteria:

* Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine), retinoids (e.g. alitretinoin) or corticosteroids within 6 weeks prior to randomization (inhaled or intra-nasal steroids corresponding to up to 1 mg prednisone for asthma or rhinitis may be used).
* PUVA (Psoralen Ultraviolet A) or UVB (Ultraviolet B) therapy on the hands within 4 weeks prior to randomization
* Cutaneously applied treatment with immunomodulators (pimecrolimus, tacrolimus) or corticosteroids on the hands within 2 weeks prior to randomization.
* Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 2 weeks prior to randomization
* Concurrent skin diseases on the hands
* Current diagnosis of exfoliative dermatitis
* Significant clinical infection (impetiginized hand eczema) on the hands which requires antibiotic treatment
* A marked abnormal ECG at baseline
* Known hepatic dysfunction or hepatic dysfunction tested at Screening
* Current participation in any other interventional clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Subjects with treatment success according to Physician's Global Assessment (PGA) at visit 6 (End of Treatment) | 56 days
  Treatment success according to the PGA is defined as: Subjects having mild disease at baseline must achieve clear. Subjects having moderate or severe disease at baseline must achieve clear or almost clear

SECONDARY OUTCOMES:
Hand Eczema Severity Index (HECSI) at visit 6 | 56 days
Subjects with treatment success according to the Patient's Global Assessment of disease severity (PaGA) at visit 6 (End of Treatment) | 56 days
  Treatment success according to the PaGA is defined as: Subjects having very mild or mild disease at baseline must achieve clear. Subjects having moderate or severe disease at baseline must achieve clear or very mild

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof Dr, Principal Investigator — Allergie-Centrum-Charité Klinik für Dermatologie, Venerologie und Allergologie
Locations (1):
- Allergie-Centrum-Charité Klinik für Dermatologie, Venerologie und Allergologie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LEO Pharma Clinical Trials — https://www.leopharmatrials.com/en